CLINICAL TRIAL: NCT03312231
Title: A Phase II Study in Healthy Adults 19 Years and Older to Assess the Safety, Reactogenicity and Immunogenicity of a Sanofi Pasteur A/H7N9 Inactivated Influenza Vaccine Administered Intramuscularly With or Without AS03 Adjuvant
Brief Title: Sanofi 2017 H7N9 With/Without AS03 in Adults/Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-0075
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Results first posted 2020-10-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2018-02-06

CONDITIONS: Avian Influenza; Influenza Immunisation
Keywords: A/H7N9; Immunogenicity; Influenza; Safety; Sanofi Pasteur; Vaccine
MeSH Terms: conditions — Influenza in Birds; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group 1 (Experimental): 3.75 mcg of H7N9 vaccine with PBS diluent plus AS03 adjuvant on days 1 and 22, n=100 (19-64 years old) and n=60 (65 and older)
  Interventions: Drug: AS03; Biological: Inactivated influenza H7N9 vaccine; Other: Phosphate Buffered Saline (PBS) diluent
- Group 2 (Experimental): 7.5 mcg of H7N9 vaccine plus AS03 adjuvant on days 1 and 22, n=100 (19-64 years old) and n=60 (65 and older)
  Interventions: Drug: AS03; Biological: Inactivated influenza H7N9 vaccine
- Group 3 (Experimental): 15 mcg of H7N9 vaccine plus AS03 adjuvant on days 1 and 22, n=100 (19-64 years old) and n=60 (65 and older)
  Interventions: Drug: AS03; Biological: Inactivated influenza H7N9 vaccine
- Group 4 (Experimental): 15 mcg of unadjuvanted H7N9 vaccine on days 1 and 22, n=50 (19-64 years old) and n=30 (65 and older)
  Interventions: Biological: Inactivated influenza H7N9 vaccine
- Group 5 (Experimental): 45 mcg of unadjuvanted H7N9 vaccine on days 1 and 22, n=50 (19-64 years old) and n=30 (65 and older)
  Interventions: Biological: Inactivated influenza H7N9 vaccine

INTERVENTIONS:
Drug: AS03 — Oil-in-water emulsion based adjuvant system.
  Arms: Group 1; Group 2; Group 3
Biological: Inactivated influenza H7N9 vaccine — Monovalent 2017 H7N9 inactivated influenza vaccine
Other: Phosphate Buffered Saline (PBS) diluent — Diluent for 2017 Monovalent Inactivated Influenza A/H7N9 virus vaccine (2017 H7N9 IIV)
  Arms: Group 1

SUMMARY:
This is a randomized, double-blinded, Phase II study in healthy males and non-pregnant females 19 years and older that is designed to assess the safety, reactogenicity, and immunogenicity of a pre-pandemic 2017 monovalent inactivated influenza A/H7N9 virus vaccine (2017 H7N9 IIV) administered at different dosages given with AS03 adjuvant and phosphate buffered saline (PBS) diluent, with AS03 adjuvant only, and without adjuvant. Eligible subjects will be randomized into 5 study groups, stratified by age. The study will enroll up to 420 individuals 19-64 years old and up to 300 individuals who are 65 years old and older. Study duration is approximately 16 months with subject participation duration approximately 13 months. The primary objectives of this study are: 1) to assess the safety and reactogenicity following receipt of two doses of 2017 H7N9 IIV administered intramuscularly at different dosages approximately 21 days apart given with or without AS03 adjuvant; 2) to assess the serum hemagglutination inhibition (HAI) and neutralizing (Neut) antibody responses following receipt of two doses of 2017 H7N9 IIV administered intramuscularly at different dosages approximately 21 days apart with or without AS03 adjuvant, stratified by age of recipient.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, Phase II study in healthy males and non-pregnant females 19 years and older. This clinical trial is designed to assess the safety, reactogenicity, and immunogenicity of a pre-pandemic 2017 monovalent inactivated influenza A/H7N9 virus vaccine (2017 H7N9 IIV) administered at different dosages given with or without adjuvant. 3.75 mcg of HA per dose will be administered with phosphate buffered saline (PBS) diluent and AS03 adjuvant, 7.5 mcg and 15 mcg of HA per dose will be administered with AS03 adjuvant only, and 15 mcg and 45 mcg of HA per dose will be administered without adjuvant. Eligible subjects will be randomized into one of 5 study groups, stratified by age. The study will enroll up to 420 individuals 19-64 years old and up to 300 individuals who are 65 years old and older. The study duration is approximately 16 months with subject participation duration approximately 13 months. The primary objectives of this study are: 1) to assess the safety and reactogenicity following receipt of two doses of 2017 H7N9 IIV administered intramuscularly at different dosages approximately 21 days apart given with or without AS03 adjuvant; 2) to assess the serum hemagglutination inhibition (HAI) and neutralizing (Neut) antibody responses following receipt of two doses of 2017 H7N9 IIV administered intramuscularly at different dosages approximately 21 days apart with or without AS03 adjuvant, stratified by age of recipient. The secondary objectives are: 1) to assess unsolicited non-serious adverse events (AEs) following receipt of two doses of a 2017 H7N9 IIV administered IM at different dosages approximately 21 days apart with or without AS03 adjuvant; 2) to assess medically-attended adverse events (MAAEs) including new-onset chronic medical conditions (NOCMCs), potentially immune-mediated medical conditions (PIMMCs), and all serious adverse events (SAEs) following receipt of two doses of a 2017 H7N9 IIV administered IM at different dosages approximately 21 days apart with or without AS03 adjuvant; 3) to assess the serum HAI and Neut antibody responses approximately 7 and 21 days following receipt of a single dose, and approximately 7 days following receipt of two doses of 2017 H7N9 IIV administered IM at different dosages approximately 21 days apart with or without AS03 adjuvant, stratified by age of recipient.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Are males or non-pregnant females, 19 years of age and older, inclusive.
4. Are in good health*. *As determined by medical history and physical examination to evaluate acute or currently ongoing chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days, which would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days (no hospitalizations, ER, or urgent care for condition and no adverse symptoms that need medical intervention such as medication change/supplemental oxygen). This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided there was no deterioration in the subject's chronic medical condition that necessitated a medication change, and there is no additional risk to the subject or interference with the evaluation of responses to study vaccination. Note: Topical, nasal, and inhaled medications (with the exception of inhaled corticosteroids as outlined in the Subject Exclusion Criteria), herbals, vitamins, and supplements are permitted.
5. Oral temperature is less than 100.0 degrees Fahrenheit.
6. Pulse is 47 to 100 bpm, inclusive.
7. Systolic blood pressure is 85 to 150 mmHg, inclusive (subjects <65 years of age), 85 to 160 mmHg, inclusive (subjects = / > 65 years of age).
8. Diastolic blood pressure is 55 to 95 mmHg, inclusive.
9. Erythrocyte sedimentation rate (ESR) is less than 30 mm per hour.
10. Women of childbearing potential* must use an acceptable contraception method** from 30 days before first study vaccination until 60 days after last study vaccination.

    *Not sterilized via tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year of the last menses if menopausal.

    **Acceptable contraception includes non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving the first study vaccination, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing(R), and licensed hormonal methods such as implants, injectables, or oral contraceptives ("the pill").
11. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to study vaccination.

Exclusion Criteria:

1. Have an acute illness*, as determined by the site principal investigator or appropriate sub-investigator, within 72 hours prior to study vaccination.

   *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site principal investigator or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
2. Have any medical disease or condition that, in the opinion of the site principal investigator or appropriate sub-investigator, is a contraindication to study participation*.

   *Including acute or chronic medical disease or condition, defined as persisting for at least 90 days, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
3. Have immunosuppression as a result of an underlying illness or treatment, a recent history or current use of immunosuppressive or immunomodulating disease therapy.
4. Use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
5. Have known active neoplastic disease or a history of any hematologic malignancy. Non-melanoma, treated, skin cancers are permitted.
6. Have known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection.
7. Have known hypersensitivity or allergy to eggs, egg or chicken protein, squalene-based adjuvants, or other components of the study vaccine.
8. Have a history of severe reactions following previous immunization with licensed or unlicensed influenza vaccines.
9. Have a personal or family history of narcolepsy.
10. Have a history of Guillain-Barré syndrome.
11. Have a history of convulsions or encephalomyelitis within 90 days prior to study vaccination.
12. Have a history of Potentially Immune-Mediated Medical Conditions (PIMMCs).
13. Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
14. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
15. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
16. Have taken oral or parenteral (including intra-articular) corticosteroids of any dose within 30 days prior to study vaccination.
17. Have taken high-dose inhaled corticosteroids* within 30 days prior to each study vaccination.

    *High-dose defined as per age as using inhaled high dose per reference chart https://www.nhlbi.nih.gov/health-pro/guidelines/current/asthma-guidelines/quick-reference-html#estimated-comparative-daily-doses
18. Received a licensed live vaccine within 30 days prior to the first study vaccination, or plan to receive a licensed live vaccine within 30 days before or after each study vaccination.
19. Received or plan to receive a licensed, inactivated, vaccine (excluding all flu vaccines) within 14 days before or after each study vaccination.
20. Received or plan to receive an inactivated seasonal flu vaccine within 21 days before or after each study vaccination.
21. Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within 90 days prior to each study vaccination.
22. Received an experimental agent* within 30 days prior to the first study vaccination, or expect to receive an experimental agent** during the 13-month trial-reporting period.

    *Including vaccine, drug, biologic, device, blood product, or medication.

    **Other than from participation in this trial.
23. Are participating or plan to participate in another clinical trial with an interventional agent* that will be received during the 13-month trial-reporting period.

    *Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.
24. Received or plan to receive an influenza A/H7 vaccine* or have a history of influenza A/H7 subtype infection.

    *And assigned to a group receiving influenza A/H7 vaccine, does not apply to documented placebo recipients.
25. Have traveled to mainland China and had substantial* direct contact with live or freshly slaughtered poultry or pigeons within the past five years.

    *Substantial contact is defined as visited a poultry farm and/or a live poultry market.
26. Occupational exposure to or substantial direct physical contact* with birds in the past year and through the 21 days after the second study vaccination.

    *Exposure to free range chickens in the yard is exclusionary. Casual contact with birds at petting zoos or county or state fairs or having pet birds does not exclude subjects from study participation.
27. Female subjects who are breastfeeding or plan to breastfeed at any given time from the first study vaccination until 30 days after the last study vaccination.
28. Plan to travel outside the US (continental US, Hawaii, and Alaska) from enrollment through 21 days after the second study vaccination.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - The Hope Clinic of Emory University, Decatur, Georgia
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - University of Maryland, School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland
  - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington

REFERENCES:
- [Derived] El Sahly HM, Anderson EJ, Jackson LA, Neuzil KM, Atmar RL, Bernstein DI, Chen WH, Creech CB, Frey SE, Goepfert P, Meier J, Phadke V, Rouphael N, Rupp R, Stapleton JT, Spearman P, Walter EB, Winokur PL, Yildirim I, Williams TL, Oshinsky J, Coughlan L, Nijhuis H, Pasetti MF, Krammer F, Stadlbauer D, Nachbagauer R, Tsong R, Wegel A, Roberts PC. Anti-neuraminidase and anti-hemagglutinin stalk responses to different influenza a(H7N9) vaccine regimens. Vaccine. 2025 Feb 15;47:126689. doi: 10.1016/j.vaccine.2024.126689. Epub 2025 Jan 4. PMID 39756216

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy males and non-pregnant females aged 19 years and older recruited from existing volunteer populations and from the communities at large around the clinical sites. Participants were enrolled between 14FEB2018 and 05SEP2018.
Groups:
- Group 1: 3.75 mcg of H7N9 vaccine plus AS03 adjuvant on days 1 and 22.
  Inactivated influenza H7N9 vaccine: Monovalent 2017 H7N9 inactivated influenza vaccine
  AS03: Oil-in-water emulsion based adjuvant system.
- Group 2: 7.5 mcg of H7N9 vaccine plus AS03 adjuvant on days 1 and 22
  Inactivated influenza H7N9 vaccine: Monovalent 2017 H7N9 inactivated influenza vaccine
  AS03: Oil-in-water emulsion based adjuvant system.
- Group 3: 15 mcg of H7N9 vaccine plus AS03 adjuvant on days 1 and 22
  Inactivated influenza H7N9 vaccine: Monovalent 2017 H7N9 inactivated influenza vaccine
  AS03: Oil-in-water emulsion based adjuvant system.
- Group 4: 15 mcg of unadjuvanted H7N9 vaccine on days 1 and 22
  Inactivated influenza H7N9 vaccine: Monovalent 2017 H7N9 inactivated influenza vaccine
- Group 5: 45 mcg of unadjuvanted H7N9 vaccine on days 1 and 22
  Inactivated influenza H7N9 vaccine: Monovalent 2017 H7N9 inactivated influenza vaccine
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Started (One subject allocated to Group 4 and received Group 5 treatment due to error was analyzed as Group 5) | 184 | 176 | 181 | 89 | 90
Completed | 181 | 165 | 177 | 86 | 89
Not Completed | 3 | 11 | 4 | 3 | 1
Not completed — Lost to Follow-up | 2 | 6 | 1 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 1 | 0 | 0
Not completed — Death | 0 | 1 | 1 | 0 | 0
Not completed — Study Vaccination not Received | 1 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all participants who received at least one dose of study vaccine.
Groups:
- Group 1: 3.75 mcg of H7N9 vaccine plus AS03 adjuvant on days 1 and 22
  Inactivated influenza H7N9 vaccine: Monovalent 2017 H7N9 inactivated influenza vaccine
  AS03: Oil-in-water emulsion based adjuvant system.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Total
Number analyzed (Participants) | 183 | 175 | 180 | 89 | 90 | 717
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (20.0) | 51.2 (20.0) | 51.5 (20.2) | 53.2 (18.6) | 51.9 (19.0) | 52.0 (19.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 99 | 81 | 47 | 50 | 371
  Male | 89 | 76 | 99 | 42 | 40 | 346
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 9 | 7 | 6 | 30
  Not Hispanic or Latino | 179 | 169 | 170 | 82 | 84 | 684
  Unknown or Not Reported | 0 | 2 | 1 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1 | 2
  Asian | 7 | 8 | 14 | 1 | 3 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 19 | 22 | 25 | 13 | 10 | 89
  White | 149 | 137 | 130 | 69 | 73 | 558
  More than one race | 6 | 5 | 7 | 4 | 2 | 24
  Unknown or Not Reported | 2 | 3 | 4 | 1 | 1 | 11
Region of Enrollment [Number; unit: participants]
  United States | 183 | 175 | 180 | 89 | 90 | 717
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.5 (5.3) | 28.2 (6.5) | 26.8 (5.4) | 27.2 (5.8) | 27.5 (4.3) | 27.5 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for HAI assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 21 days after the second dose of H7N9.
Time Frame: Day 43
Population: The modified intent-to-treat (mITT) population includes all participants who received at least one study vaccination and contributed both pre- and at least one post-study vaccination venous blood samples for HAI antibody assays for which valid results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 179 | 172 | 180 | 87 | 88
titer | 33.6 [27.8 to 40.7] | 33.5 [27.9 to 40.2] | 39.2 [32.6 to 47.0] | 5.5 [5.3 to 5.7] | 6.3 [5.7 to 6.9]

2. Primary Outcome: Geometric Mean Titers (GMTs) of Serum Neutralizing (Neut) Antibodies
Description: Blood was collected for Neutralizing assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 21 days after the second dose of H7N9.
Time Frame: Day 43
Population: The modified intent-to-treat (mITT) population includes all participants who received at least one study vaccination and contributed both pre- and at least one post-study vaccination venous blood samples for Neut antibody assays for which valid results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 179 | 173 | 180 | 87 | 88
titer | 45.2 [38.4 to 53.2] | 46.1 [39.5 to 53.9] | 49.7 [42.5 to 58.1] | 6.2 [5.7 to 6.8] | 7.8 [6.8 to 9.0]

3. Primary Outcome: Number of Participants With Clinical Safety Laboratory Adverse Events
Description: Laboratory parameters include alanine aminotransferase (ALT), bilirubin, creatinine, hemoglobin, platelets and white blood cells (WBC). Thresholds for adverse events were considered as ALT 44 IU/L or greater (female) or 61 IU/L or greater (male); bilirubin 1.30 mg/dL or greater; creatinine 1.1 mg/dL or greater (female) or 1.4 mg/dL or greater (male); hemoglobin 11.4 g/dL or lower (female) or 12.4 g/dL or lower (male); platelets 139 x10^3/µL or below or 416 x10^3/µL or greater; or WBC or 3.9 x10^3/µL or lower or 10.6 x10^3/µL or higher.
Time Frame: Day 8
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine. Participants who completed Day 8 visit were included for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 182 | 173 | 179 | 88 | 90
Participants
  WBC | 8 | 18 | 16 | 6 | 5
  Hemoglobin | 4 | 5 | 3 | 8 | 5
  Platelets | 4 | 7 | 1 | 2 | 3
  ALT | 3 | 5 | 3 | 1 | 1
  Total Bilirubin | 0 | 3 | 2 | 4 | 1
  Creatinine | 2 | 5 | 4 | 2 | 3

4. Primary Outcome: Number of Participants With Clinical Safety Laboratory Adverse Events
Description: as for outcome 3
Time Frame: Day 29
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine. Participants who completed Day 29 visit were included for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 169 | 156 | 169 | 83 | 78
Participants
  WBC | 10 | 14 | 14 | 7 | 4
  Hemoglobin | 7 | 8 | 5 | 6 | 3
  Platelets | 3 | 2 | 2 | 1 | 3
  ALT | 2 | 3 | 2 | 1 | 0
  Total Bilirubin | 2 | 5 | 2 | 0 | 1
  Creatinine | 2 | 4 | 3 | 2 | 3

5. Primary Outcome: Number of Participants Reporting Solicited Injection Site Events
Description: Injection site AEs solicited on a memory aid provided to participants included Pain, Tenderness, Itching/Pruritus, Ecchymosis/Bruising (functional grade based on interference with dailyactivities), Ecchymosis/Bruising (any measured value >0mm), Erythema/Redness (functional grade), Erythema/ Redness (any measured value >0mm), Induration/Swelling (functional grade), and Induration/Swelling (any measured value >0mm). Participants are considered reporting the injection site AE if they reported mild or greater severity at any time during the 8 days at or following the first vaccination.
Time Frame: Day 1 to Day 8
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 175 | 180 | 89 | 90
Participants | 145 | 153 | 154 | 36 | 46

6. Primary Outcome: Number of Participants Reporting Solicited Injection Site Events
Description: Injection site AEs solicited on a memory aid provided to participants included Pain, Tenderness, Itching/Pruritus, Ecchymosis/Bruising (functional grade based on interference with dailyactivities), Ecchymosis/Bruising (any measured value >0mm), Erythema/Redness (functional grade), Erythema/ Redness (any measured value >0mm), Induration/Swelling (functional grade), and Induration/Swelling (any measured value >0mm). Participants are considered reporting the injection site AE if they reported mild or greater severity at any time during the 8 days at or following the second vaccination.
Time Frame: Day 22 to Day 29
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 173 | 157 | 170 | 84 | 78
Participants | 122 | 116 | 140 | 35 | 33

7. Primary Outcome: Number of Participants Reporting Study Vaccine-related Serious Adverse Events (SAEs)
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect. Events are included if deemed by the investigator to be related to the study product.
Time Frame: Day 1 to Day 387
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 175 | 180 | 89 | 90
Participants | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Events
Description: Systemic AEs solicited on a memory aid provided to participants included Elevated Oral Temperature, Feverishness, Fatigue, Malaise, Myalgia, Arthralgia, Headache, and Nausea. Participants are considered reporting the systemic AE if they reported mild or greater severity at any time during the 8 days at or following the first vaccination.
Time Frame: Day 1 to Day 8
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 175 | 180 | 89 | 90
Participants | 76 | 81 | 72 | 27 | 31

9. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Events
Description: Systemic AEs solicited on a memory aid provided to participants included Elevated Oral Temperature, Feverishness, Fatigue, Malaise, Myalgia, Arthralgia, Headache, and Nausea. Participants are considered reporting the systemic AE if they reported mild or greater severity at any time during the 8 days at or following the second vaccination.
Time Frame: Day 22 to Day 29
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 173 | 157 | 170 | 84 | 78
Participants | 75 | 64 | 72 | 19 | 17

10. Primary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibodies Titer of 1:40 or Greater
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study group from the available results at 21 days after second dose of H7N9.
Time Frame: Day 43
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 179 | 172 | 180 | 87 | 88
percentage of participants | 57 [49 to 64] | 56 [49 to 64] | 61 [54 to 68] | 0 [0 to 4] | 2 [0 to 8]

11. Primary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibodies Titer of 1:40 or Greater
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study group from the available results at 21 days after second dose of H7N9.
Time Frame: Day 43
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 179 | 173 | 180 | 87 | 88
proportion of participants | 64 [56 to 71] | 65 [57 to 72] | 68 [60 to 75] | 0 [0 to 4] | 3 [1 to 10]

12. Primary Outcome: Percentage of Participants Achieving Seroconversion Defined by Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >=1:40 or pre-vaccination titer 1:10 or greater and minimum 4-fold rise in post-vaccination antibody titer. 21 days after second dose of H7N9 is Day 43.
Time Frame: Day 43
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 179 | 172 | 180 | 87 | 88
percentage of participants | 56 [49 to 64] | 56 [49 to 64] | 61 [54 to 68] | 0 [0 to 4] | 2 [0 to 8]

13. Primary Outcome: Percentage of Participants Achieving Seroconversion Defined by Neutralizing (Neut) Antibodies
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >=1:40 or pre-vaccination titer 1:10 or greater and minimum 4-fold rise in post-vaccination antibody titer. 21 days after second dose of H7N9 is Day 43.
Time Frame: Day 43
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 179 | 173 | 180 | 87 | 88
percentage of participants | 64 [56 to 71] | 64 [56 to 71] | 67 [60 to 74] | 0 [0 to 4] | 2 [0 to 8]

14. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for HAI assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at baseline.
Time Frame: Day 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 174 | 180 | 88 | 90
titer | 5.2 [5.1 to 5.3] | 5.2 [5.1 to 5.3] | 5.2 [5.1 to 5.3] | 5.3 [5.1 to 5.4] | 5.4 [5.1 to 5.6]

15. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for HAI assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 7 days post first vaccination.
Time Frame: Day 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 173 | 180 | 88 | 90
titer | 5.3 [5.1 to 5.5] | 5.6 [5.2 to 6.1] | 5.8 [5.5 to 6.2] | 5.3 [5.1 to 5.5] | 6.0 [5.2 to 6.9]

16. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for HAI assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 21 days post first vaccination.
Time Frame: Day 22
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 182 | 173 | 179 | 87 | 90
titer | 6.7 [6.2 to 7.3] | 7.0 [6.4 to 7.7] | 7.6 [6.9 to 8.5] | 5.5 [5.2 to 5.9] | 6.0 [5.2 to 6.9]

17. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for HAI assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 7 days post second vaccination.
Time Frame: Day 29
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 171 | 155 | 170 | 83 | 78
titer | 36.7 [29.9 to 45.2] | 45.1 [37.1 to 54.9] | 45.7 [37.6 to 55.5] | 5.4 [5.2 to 5.6] | 6.8 [6.0 to 7.7]

18. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Neutralizing (Neut) Antibodies
Description: Blood was collected for Neutralizing assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at baseline.
Time Frame: Day 1
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 174 | 180 | 88 | 90
titer | 5.2 [5.1 to 5.4] | 5.3 [5.1 to 5.5] | 5.3 [5.2 to 5.5] | 5.3 [5.1 to 5.6] | 5.5 [5.1 to 6.0]

19. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Neutralizing (Neut) Antibodies
Description: Blood was collected for Neutralizing assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 7 days post first vaccination.
Time Frame: Day 8
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 173 | 180 | 88 | 90
titer | 5.6 [5.4 to 5.8] | 6.4 [5.8 to 7.0] | 6.6 [6.1 to 7.1] | 5.5 [5.2 to 5.8] | 6.3 [5.5 to 7.3]

20. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Neutralizing (Neut) Antibodies
Description: Blood was collected for Neutralizing assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 21 days post first vaccination.
Time Frame: Day 22
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 182 | 172 | 179 | 87 | 90
titer | 8.4 [7.7 to 9.2] | 9.1 [8.1 to 10.2] | 9.9 [8.8 to 11.1] | 5.4 [5.2 to 5.6] | 6.9 [5.9 to 8.0]

21. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Neutralizing (Neut) Antibodies
Description: Blood was collected for Neutralizing assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm from the available results at 7 days post second vaccination.
Time Frame: Day 29
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 172 | 156 | 168 | 83 | 78
titer | 43.6 [36.5 to 52.2] | 53.9 [45.6 to 63.6] | 54.7 [46.1 to 64.9] | 6.1 [5.6 to 6.6] | 8.1 [6.9 to 9.5]

22. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs), Regardless of the Assessment of Relatedness
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect. All events are included regardless of relationship to the study product.
Time Frame: Day 1 to Day 387
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 175 | 180 | 89 | 90
Participants | 4 | 9 | 4 | 3 | 1

23. Secondary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs), Regardless of the Assessment of Seriousness or Relatedness
Description: Adverse events were defined as any untoward medical occurrence in a participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Non-serious AEs were collected from participants at follow up visits through 21 days after each vaccination. Adverse events were MedDRA coded and are summarized by MedDRA System Organ Class (SOC).
Time Frame: Day 1 to Day 43
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 175 | 180 | 89 | 90
Participants | 72 | 62 | 67 | 23 | 27

24. Secondary Outcome: Number of Participants Reporting Medically-attended Adverse Events (MAAEs), New-onset Chronic Medical Conditions (NOCMCs), and Potentially Immune-mediated Medical Conditions (PIMMCs)
Description: For each unsolicited AE experienced, the participants were asked if he/she had received medical attention, defined as hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel for any reason. AEs characterized by such unscheduled medical care were designated as MAAEs. NOCMCs are defined as any new ICD-10 diagnosis that is applied to the participant during the duration of the study, after receipt of the study agent, that is expected to continue for at least 3 months and requires continued health care intervention. PIMMCs constitute a group of AEs that includes diseases which are clearly autoimmune in etiology and other inflammatory and/or neurologic disorders which may or may not have autoimmune etiologies.
Time Frame: Day 1 to Day 387
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 175 | 180 | 89 | 90
Participants
  Medically-Attended Adverse Events | 69 | 59 | 65 | 33 | 25
  New-Onset Chronic Medical Conditions | 17 | 7 | 7 | 7 | 4
  Potentially Immune-Mediated Medical Conditions | 2 | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Participants Reporting Study Vaccine-related Unsolicited Non-serious Adverse Events (AEs)
Description: Adverse events were defined as any untoward medical occurrence in a participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Non-serious AEs were collected from participants at follow up visits through 21 days after each vaccination. The site investigator determined vaccine related as "a reasonable possibility that the study product caused the AE. Reasonable possibility means that there is evidence to suggest a causal relationship between the study product and the AE." Adverse events were MedDRA coded and are summarized by MedDRA System Organ Class (SOC).
Time Frame: Day 1 to Day 43
Population: The Safety Analysis population includes all participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 175 | 180 | 89 | 90
Participants | 19 | 14 | 12 | 4 | 4

26. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibodies Titers of 1:40 or Greater
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study group from the available results at baseline.
Time Frame: Day 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 174 | 180 | 88 | 90
percentage of participants | 0 [0 to 2] | 0 [0 to 2] | 0 [0 to 2] | 0 [0 to 4] | 0 [0 to 4]

27. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibodies Titers of 1:40 or Greater
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study group from the available results at 7 days post first vaccination.
Time Frame: Day 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 173 | 180 | 88 | 90
percentage of participants | 1 [0 to 3] | 2 [0 to 5] | 2 [1 to 6] | 0 [0 to 4] | 2 [0 to 8]

28. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibodies Titers of 1:40 or Greater
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study group from the available results at 21 days post first vaccination.
Time Frame: Day 22
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 182 | 173 | 179 | 87 | 90
percentage of participants | 3 [1 to 7] | 5 [2 to 10] | 7 [4 to 11] | 1 [0 to 6] | 2 [0 to 8]

29. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibodies Titers of 1:40 or Greater
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study group from the available results at 7 days post second vaccination.
Time Frame: Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 171 | 155 | 170 | 83 | 78
percentage of participants | 57 [49 to 64] | 65 [57 to 73] | 64 [56 to 71] | 0 [0 to 4] | 5 [1 to 13]

30. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibodies Titers of 1:40 or Greater
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study group from the available results at baseline.
Time Frame: Day 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 174 | 180 | 88 | 90
percentage of participants | 0 [0 to 2] | 1 [0 to 3] | 0 [0 to 2] | 0 [0 to 4] | 1 [0 to 6]

31. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibodies Titers of 1:40 or Greater
Description: as for outcome 27
Time Frame: Day 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 173 | 180 | 88 | 90
percentage of participants | 0 [0 to 2] | 3 [1 to 7] | 2 [0 to 5] | 0 [0 to 4] | 3 [1 to 9]

32. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibodies Titers of 1:40 or Greater
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study group from the available results at 21 days post first vaccination.
Time Frame: Day 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 182 | 172 | 179 | 87 | 90
percentage of participants | 2 [1 to 6] | 5 [2 to 10] | 6 [3 to 11] | 0 [0 to 4] | 3 [1 to 9]

33. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibodies Titers of 1:40 or Greater
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study group from the available results at 7 days post second vaccination.
Time Frame: Day 29
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 172 | 156 | 168 | 83 | 78
percentage of participants | 61 [53 to 68] | 71 [63 to 78] | 67 [60 to 74] | 0 [0 to 4] | 6 [2 to 14]

34. Secondary Outcome: Percentage of Participants Achieving Seroconversion Defined by Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >=1:40 or pre-vaccination titer 1:10 or greater and minimum 4-fold rise in post-vaccination antibody titer. Day 8 is 7 days after the first dose of H7N9.
Time Frame: Day 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 173 | 180 | 88 | 90
percentage of participants | 0 [0 to 2] | 1 [0 to 4] | 2 [1 to 6] | 0 [0 to 4] | 2 [0 to 8]

35. Secondary Outcome: Percentage of Participants Achieving Seroconversion Defined by Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >=1:40 or pre-vaccination titer 1:10 or greater and minimum 4-fold rise in post-vaccination antibody titer. Day 22 is 21 days after the first dose of H7N9.
Time Frame: Day 22
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 182 | 173 | 179 | 87 | 90
percentage of participants | 3 [1 to 6] | 5 [2 to 10] | 7 [4 to 11] | 1 [0 to 6] | 2 [0 to 8]

36. Secondary Outcome: Percentage of Participants Achieving Seroconversion Defined by Hemagglutination Inhibition (HAI) Antibodies
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >=1:40 or pre-vaccination titer 1:10 or greater and minimum 4-fold rise in post-vaccination antibody titer. Day 29 is 7 days after the second dose of H7N9.
Time Frame: Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 171 | 155 | 170 | 83 | 78
percentage of participants | 56 [48 to 64] | 65 [57 to 73] | 64 [56 to 71] | 0 [0 to 4] | 5 [1 to 13]

37. Secondary Outcome: Percentage of Participants Achieving Seroconversion Defined by Neutralizing (Neut) Antibodies
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >=1:40 or pre-vaccination titer 1:10 or greater and minimum 4-fold rise in post-vaccination antibody titer. Day 8 is 7 days after the first dose of H7N9.
Time Frame: Day 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 183 | 173 | 180 | 88 | 90
percentage of participants | 0 [0 to 2] | 2 [1 to 6] | 2 [0 to 5] | 0 [0 to 4] | 2 [0 to 8]

38. Secondary Outcome: Percentage of Participants Achieving Seroconversion Defined by Neutralizing (Neut) Antibodies
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >=1:40 or pre-vaccination titer 1:10 or greater and minimum 4-fold rise in post-vaccination antibody titer. Day 22 is 21 days after the first dose of H7N9.
Time Frame: Day 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 182 | 172 | 179 | 87 | 90
percentage of participants | 2 [0 to 5] | 5 [2 to 9] | 6 [3 to 11] | 0 [0 to 4] | 2 [0 to 8]

39. Secondary Outcome: Percentage of Participants Achieving Seroconversion Defined by Neutralizing (Neut) Antibodies
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >=1:40 or pre-vaccination titer 1:10 or greater and minimum 4-fold rise in post-vaccination antibody titer. Day 29 is 7 days after the second dose of H7N9.
Time Frame: Day 29
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
Number analyzed (Participants) | 172 | 156 | 168 | 83 | 78
percentage of participants | 60 [53 to 68] | 70 [62 to 77] | 67 [59 to 74] | 0 [0 to 4] | 6 [2 to 14]

ADVERSE EVENTS:
Time Frame: Solicited events were collected from the time of each study vaccination through 7 days after each study vaccination. Unsolicited non-serious AEs were collected from the time of each study vaccination through approximately 21 days after each study vaccination. SAEs and MAAEs, including NOCMCs and PIMMCs, were collected from the time of the first study vaccination through the final study visit, approximately 12 months after the last study vaccination.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Group 5
All-Cause Mortality (participants affected / at risk) | 1/183 | 1/175 | 1/180 | 0/89 | 0/90
Serious Adverse Events (participants affected / at risk) | 4/183 | 9/175 | 4/180 | 3/89 | 1/90
Other Adverse Events (participants affected / at risk) | 172/183 | 170/175 | 167/180 | 70/89 | 73/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=183) | Group 2 (N=175) | Group 3 (N=180) | Group 4 (N=89) | Group 5 (N=90)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=183) | Group 2 (N=175) | Group 3 (N=180) | Group 4 (N=89) | Group 5 (N=90)
Nausea (Gastrointestinal disorders) | 18 (18) | 19 (21) | 13 (14) | 3 (3) | 4 (4)
Fatigue (General disorders) | 65 (86) | 67 (82) | 67 (94) | 21 (25) | 21 (24)
Feverishness (General disorders) | 28 (34) | 31 (35) | 35 (41) | 1 (1) | 6 (7)
Injection site pruritus (General disorders) | 19 (22) | 12 (12) | 14 (17) | 2 (2) | 4 (4)
Injection site erythema (General disorders) | 51 (61) | 47 (58) | 58 (76) | 23 (30) | 25 (31)
Injection site haemorrhage (General disorders) | 17 (18) | 22 (23) | 18 (21) | 3 (3) | 10 (11)
Injection site induration (General disorders) | 46 (54) | 41 (52) | 62 (84) | 11 (11) | 14 (15)
Injection site pain (General disorders) | 87 (128) | 99 (140) | 110 (170) | 12 (15) | 15 (18)
Injection site tenderness (General disorders) | 142 (233) | 146 (230) | 150 (258) | 28 (41) | 37 (46)
Malaise (General disorders) | 45 (51) | 44 (53) | 44 (56) | 5 (5) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 10 (12) | 14 (16) | 6 (7) | 6 (6)
Haemoglobin decreased (Investigations) | 9 (18) | 12 (23) | 5 (12) | 11 (23) | 7 (12)
Platelet count decreased (Investigations) | 2 (5) | 5 (9) | 3 (3) | 2 (3) | 5 (8)
White blood cell count decreased (Investigations) | 20 (29) | 18 (28) | 24 (42) | 13 (18) | 10 (17)
White blood cell count increased (Investigations) | 1 (3) | 9 (12) | 1 (2) | 4 (6) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 (35) | 21 (23) | 35 (38) | 7 (9) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 57 (74) | 57 (68) | 57 (75) | 10 (13) | 16 (18)
Headache (Nervous system disorders) | 55 (66) | 51 (60) | 52 (61) | 19 (21) | 18 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT03312231/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT03312231/SAP_001.pdf